CLINICAL TRIAL: NCT05253235
Title: Can Family-Centered Prevention Programming Reduce Neuroimmune Vulnerabilities for Drug Use and Cardiometabolic Risk Among African American Adolescents? A Randomized Prevention Trial
Brief Title: Health and Resilience Projects: Foundations
Acronym: HARP-F
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Gene H. Brody, Regents Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PROJECT00003530
Record Dates: First submitted 2022-02-01; First posted 2022-02-23 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to a preventive intervention or a no treatment control
Who Masked: Outcomes Assessor
Masking Description: Assessment staff will be blind to families' experimental assignment at pretest.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAAF Intervention (Experimental): Parents and youth will receive an online, family-centered intervention consisting of 7 weekly sessions.
  Interventions: Behavioral: SAAF
- Control Group (Other): Control group members will receive a book entitled, Parenting for Liberation: A Guide for Raising Black Children
  Interventions: Other: Receipt of parenting book

INTERVENTIONS:
Behavioral: SAAF — A 7 session online intervention designed to augment protective processes associated with deterrence of substance use
  Arms: SAAF Intervention
Other: Receipt of parenting book — Parents will receive a copy of the book, Parenting for Liberation: A Guide for Raising Black Children
  Arms: Control Group

SUMMARY:
The Health and Resilience Project (HARP): Foundations is investigating the efficacy of the Strong African American Families (SAAF) intervention in promoting the health and well being of African American adolescents. Youth age 10-13 and their primary caregivers are randomly assigned to receive SAAF or to a control group. Participants complete baseline and follow-up measures regarding vulnerability to substance use based on a neuroimmune model of stress coping.

DETAILED DESCRIPTION:
During childhood and adolescence, family relationships play critical roles in regulating physiological stress reactions. This protects the developing brain from the potentially deleterious effects of stress hormones and neurochemicals. In a series of proof-of-principle studies, the investigators studied the potential for the Strong African American Families (SAAF) drug use prevention program delivered when youth were age 11 to protect participants from the consequences of social adversity when they were transitioning to adulthood (ages 19-25). Effects were detected on a range of outcomes associated with neuroimmune (NIN) dysregulation including inflammation, the neural structure of limbic regions, prefrontal-limbic connectivity, and cardiometabolic health. Although these findings are provocative, the SAAF trial was not designed to evaluate mechanisms and outcomes that the NIN model suggested. Data on inflammation and neural activity were collected post hoc, many years after the intervention concluded. Thus these findings must be regarded as preliminary until a more rigorous study is performed with pretest and posttest measures of NIN processes. The proposed prevention trial of SAAF (N = 325) is designed to meet this need.

Our specific aims are to test hypotheses regarding:

1. the influence of participation in SAAF on change in NIN-associated risk markers (neural circuitry subserving threat, reward, and executive control, as well as peripheral inflammation) across 2 years;
2. the mediating role of protective parenting in linking intervention participation to NIN-associated risk markers;
3. the influence of participation in SAAF on change in addictive behavior vulnerabilities associated with risky decision making, emotion regulation, early-onset substance use, unhealthy eating, and cardiometabolic risk markers; and
4. the mediational chain linking SAAF to addictive behavior vulnerabilities via changes in parenting and NIN-associated risk markers.

A sample of 325 African American youth and their primary caregivers will be recruited from Athens, GA and surrounding areas. Inclusion criteria are (a) youth or parent self-designates as African American, Black, or biracial (including Black or African American), and (b) youth is in 5th grade and 10-13 years of age. Exclusion criteria include: (a) contraindications for MRI scanning (e.g., metal in body, traumatic brain injury, claustrophobia, pregnancy), (b) youth with chronic illnesses or medication regimens that would affect inflammatory panels (e.g., diabetes, congenital heart disease, asthma, cancers), and (c) parent or youth conditions (e.g., ADHD, psychoses) that would prevent participation in the SAAF intervention. Given the nonverbal nature of fMRI tasks, left-handed youth are not excluded. The investigators anticipate screening ~615 families over a 2.5-year period to obtain a sample of 325 families. Eligible participants will be scheduled for an assessment at UGA's Bioimaging Research Center. Youth will participate in a scan (~60 minutes), a blood draw, and youth and parents will complete self-report measures. At each data collection wave, parents consent in writing to their own and their children's participation and children provide written assent. At W2, a home visit is made with laptop computers to collect self-report data. After pretest, families will be assigned randomly to SAAF or control. Control families receive written information by mail regarding adolescent development.

ELIGIBILITY:
Inclusion Criteria:

Youth:

* Self reported African American or Black;
* Age 10-13

Parents:

* Primary caregiver for youth,
* Resides in same household as youth.

Exclusion Criteria:

Youth :

* Contraindications for MRI scanning (e.g., metal in body, traumatic brain injury, claustrophobia, pregnancy),
* Youth with chronic illnesses or medication regimens that would affect inflammatory panels (e.g., diabetes, congenital heart disease, asthma, cancers).

Parent:

* Conditions (e.g., severe disability, psychoses) that would prevent participation in the SAAF intervention or completing self-report measures.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 650 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-regulation (youth report) | Two years
  Youth will complete the the Future-oriented Goals scale and Will's Self-Control scale. We will standardize scores from these two measures (mean =0, standard deviation =1) then average them together. We expect assignment to SAAF vs control to be associated with higher scores (more self-regulation).
Self-regulation (parent report) | Two years
  Parents will complete a 12 item scale (Humphrey's self control scale) about their youth. Items will be summed ranging from 0-36. We expect assignment to SAAF vs control to be associated with higher scores (more self-regulation).
Tolerance for Deviance Scale | Two years
  Youth will complete the Tolerance for Deviance scale. 19 Items are summed, ranging from 0-57. We expect assignment to SAAF vs Control to be associated with lower scores (reductions in risky attitudes).
Reward-based eating | Two years
  Youth will complete the 13 items Reward Based Eating Drive scale. Scores range from 13-65. SAAF youth are expected to have lower scores on reward based eating compared to control youth.
Substance use onset | Two years
  Lifetime use (yes or no) of alcohol, marijuana, or cigarettes per youth self-report. We will sum the items to form a composite onset index. We expect youth assigned to SAAF to report less substance use onset than youth assigned to control.
Past 3 month substance use frequency | Two years
  Youth complete likert type items assessing alcohol, marijuana, and nicotine use in the past 3 months. Items are standardized and summed to form a substance use composite. We expect youth assigned to SAAF to report less substance use than youth assigned to control.
Unhealthy eating | Two Years
  Youth will complete the Adolescent Food Habits checklist. Items are summed. We expect SAAF youth to engage in less unhealthy eating than control youth.

SECONDARY OUTCOMES:
Involved Vigilant Parenting Scale (youth report) | 1 year
  Youth report on the 17 item Involved Vigilant Parenting scale. Items are summed to indicate higher scores on effective parenting, ranging from 17-85. We expect SAAF youth to report more involved vigilant parenting than control youth.
Involved Vigilant Parenting (parent report) | 1 year
  Parents report on the 17 item Involved Vigilant Parenting scale. Items are summed to indicate higher scores on effective parenting, ranging from 17-85. We expect SAAF parents to report more involved vigilant parenting than control parents.
Cultural socialization (youth report) | 1 year
  Youth report on the cultural socialization subscale of the Racial Socialization Scale. Five items (range is 5-25) are summed to indicate higher scores on cultural socialization. We expect SAAF youth to report more cultural socialization than control youth.
Cultural socialization (parent report) | 1 year
  Caregivers report on the cultural socialization subscale of the Racial Socialization Scale. Five items (range is 5-25) are summed to indicate higher scores on cultural socialization. We expect SAAF parents to report more cultural socialization than control parents.
Communication about Risk Behavior (youth report) | 1 year
  Youth report on Discussion Quality scale. Three items are summed to indicate higher scores on communication (range 0-12). We expect SAAF youth to report more harmonious communication than control youth.
Communication about risk behavior (parent report) | 1 year
  Parents report on the Discussion Quality scale. Three items are summed to indicate higher scores on communication (range 0-12). We expect SAAF parents to report more harmonious communication than control parents.
Threat sensitivity via functional MRI assessment | Two years
  Threat sensitivity is assessed via amygdalar activity during a threat paradigm. We expect assignment to SAAF to be associated with diminished amygdalar reactivity to threat stimuli.
Executive control assessed via functional MRI assessment | Two years
  We will use multivariate autoregressive modeling to generate parameter estimates of functional connectivity within cortico-amygdalar and cortico-striatal circuitry during the reward task. We focus on a seed-to-seed association between the orbital frontal cortext (OFC) and the ventral striatum (VS). Here, a positive (i.e., > 0) parameter estimate reflects strong executive control over the VS during reward processing. Conversely, a negative parameter estimate (i.e., < 0) suggests the youth is engaging the OFC in a manner that down-regulates sub-cortical reward processing.
Reward sensitivity via functional MRI assessment | Two years
  Neural activity associated with processing rewarding stimuli using fMRI data. We predict that assignment to SAAF will reduce deficits in reward sensitivity as assessed by ventral striatum activity during a reward task.
Peripheral inflammation composite score | Two years
  Inflammatory signaling is assessed via a composite measure of circulating cytokines (Interleukin [IL]-6, 8, 10, tumor necrosis factor [TNF]-α) and C-reactive protein (CRP). Per past research, we will standardize the values for each biomarker and then sum them to form a composite score ranging from 0-5. A higher score on this composite reflects more low-grade inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Gene H Brody, Ph.D., Principal Investigator — University of Georgia
Locations (1):
- Center for Family Research, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in a specific article, after deidentification (text, tables, figures, and appendices), will be made available to qualified researchers, beginning 9 months after publication and ending 36 months after publication. Data will be shared with investigators whose proposed use of the data has been approved by a review committee designated for this purpose. Proposals should be directed to Gene Brody gbrody@uga.edu. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP
Time Frame: Available 9 months to 36 months after article publication
Access Criteria: Investigators working under an institution with a Federal Wide Assurance (FWA) and have received approval from a certified Institutional Review Board may request data.